CLINICAL TRIAL: NCT06686927
Title: Study on Glucocorticoid Combined With Gamma Globulin and Ropristine N01 in Treatment of Initial Severe ITP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0503
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-08

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: severe ITP; Romiplostim
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins; romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corticosteroids combined with immunoglobulin and romiplostim (Experimental): Romiplostim N01, starting dose of 1 µg/kg, subcutaneous injection, given on the third day of IVIG, once a week, for up to one month.
  IVIG, 400mg/kg/d, intravenous administration, continuous administration for 3-5 days.
  Prednisone, 0.8mg/kg/d, taken orally or intravenously, for up to one month.
  Interventions: Drug: corticosteroids combined with immunoglobulin and romiplostim

INTERVENTIONS:
Drug: corticosteroids combined with immunoglobulin and romiplostim — Romiplostim N01, starting dose of 1 µg/kg, subcutaneous injection, given on the third day of IVIG, once a week, for up to one month.
  IVIG, 400mg/kg/d, intravenous administration, continuous administration for 3-5 days.
  Prednisone, 0.8mg/kg/d, taken orally or intravenously, for up to one month.

SUMMARY:
The goal of this clinical trial is to learn if romiplostim N01 works to treat severe primary immune thrombocytopenia in adults. It will also learn about the safety of romiplostim N01. The main question it aims to answer is:

TO evaluate the effectiveness of the combination treatment of glucocorticoids, gamma globulin and romiplostim N01 in patients with severe primary immune thrombocytopenia during the initial treatment period for one month.

Participants will:

Romiplostim N01, starting dose of 1 µg/kg, subcutaneous injection, given on the third day of IVIG, once a week, for up to one month.

IVIG, 400mg/kg/d, intravenous administration, continuous administration for 3-5 days.

Prednisone, 0.8mg/kg/d, taken orally or intravenously, for up to one month.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign a written informed consent prior to enrollment;
2. Ages 18-75;
3. Platelet count <10×10^9/L with active bleeding or bleeding score ≥5;
4. No contraindications to the use of steroids, romiplostim, or IVIG, and willingness to receive these treatments;
5. No prior splenectomy or at least one first-line ITP treatment or emergency treatment;
6. No prior romiplostim treatment;
7. ECOG PS score: 0-2;
8. Female participants of childbearing potential must agree to use reliable contraception (including male or female condoms, contraceptive foam, contraceptive jelly, contraceptive patches, contraceptive cream, contraceptive suppositories, abstinence, and placement of intrauterine contraceptive devices) throughout the study; women who have had a hysterectomy, bilateral oophorectomy, bilateral salpingo-oophorectomy, or have been postmenopausal for more than 1 year, and men who have had bilateral vasectomy or vasectomy are excluded;
9. Voluntary participation in this study and good compliance.

Exclusion Criteria:

1. Individuals with the following hematological disorders other than ITP, including but not limited to leukemia, thrombocytopenia caused by cancer treatment, myeloproliferative diseases, multiple myeloma, and myelodysplastic syndrome;
2. Individuals with a history of thrombosis;
3. Pregnant or lactating individuals;
4. Individuals with severe cardiopulmonary insufficiency;
5. Individuals with severe or uncontrollable infections;
6. Individuals with viral infections;
7. Individuals who cannot comply due to psychological reasons;
8. Individuals who are deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The total effective rate of treatment for 30 days | one months
  GR = CR + R (Complete reaction CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Effective R, platelet count between 30×10^9/L and 100×10^9/L, and at least double the baseline value, and no bleeding symptoms)

SECONDARY OUTCOMES:
Early (week) response rate R | one months
  Effective R, platelet count between 30×10^9/L and 100×10^9/L, and at least double the baseline value, and no bleeding symptoms
Early Complete Response Rate (CR) | one months
  Complete reaction CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms
Time to Reaction | one months
  Time of Starting Treatment Until Platelet Count ≥ 30×10^9/L
Adverse events during treatment | four months
  evaluated using Version 5.0 of the "Common Terminology Criteria for Adverse Events(NCI CTC AE)"

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No